CLINICAL TRIAL: NCT03652610
Title: Immunogenicity, Reactogenicity and Safety of Two Formulations of GSK Biologicals' Meningococcal ACWY Conjugate Vaccine (GSK3536820A and Menveo) in Healthy Adults 18 to 40 Years of Age
Brief Title: A Study to Investigate the Safety and Immunogenicity of Different Formulations of GSK Biologicals' Meningococcal ACWY Conjugate Vaccine (GSK3536820A and Menveo) Administered to Healthy Adults 18 to 40 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205343; V59_71 (Other: Novartis); 2017-003692-61 (EudraCT Number)
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Infections, Meningococcal
Keywords: Meningitis; Liquid formulation; Meningococcal disease
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner. By observer-blind, it is meant that during the course of the study, the vaccine recipient and those responsible for the evaluation of any study endpoint (e.g. safety, reactogenicity and immunogenicity) will all be unaware of which vaccine was administered. To do so, vaccine preparation and administration will be done by authorized medical personnel who will not participate in any of the study clinical evaluations.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK3536820A ACWY_Liq Group (Experimental): Healthy adults, 18 to 40 years of age, receiving at Day 1 a single dose of investigational MenACWY liquid vaccine (GSK3536820A) formulation with approximately 30% Men A FS.
  Interventions: Biological: MenACWY liquid vaccine with approximately 30% MenA FS (GSK3536820A)
- ACWY Group (Active Comparator): Healthy adults 18 to 40 years of age, receiving at Day 1 a single dose of licensed GSK's MenACWY vaccine formulation (Menveo).
  Interventions: Biological: Licensed GSK MenACWY vaccine (Menveo)

INTERVENTIONS:
Biological: MenACWY liquid vaccine with approximately 30% MenA FS (GSK3536820A) — Single dose administered at Day 1, by intramuscular injection in the deltoid of the non-dominant arm
  Other Names: GSK3536820A
  Arms: GSK3536820A ACWY_Liq Group
Biological: Licensed GSK MenACWY vaccine (Menveo) — Single dose administered at Day 1, by intramuscular injection in the deltoid of the non-dominant arm
  Arms: ACWY Group

SUMMARY:
MenACWY (Menveo) is a GSK vaccine intended for protection against disease caused by meningococcal bacteria groups A, C, W and Y in infants, children and adults, licensed in more than 60 countries.

The purpose of this study is to compare the immunogenicity of the currently licensed MenACWY vaccine with the investigational MenACWY liquid vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol or subjects' parent(s)/Legally Acceptable Respresentative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
2. Written informed consent obtained from the subject/from the parents(s)/LAR(s) of the subject prior to performance of any study specific procedure.
3. Written informed assent obtained for subjects below legal age of consent, if required by local regulations, at the time of enrolment.
4. A male or female between, and including, ≥18 to ≤40 YoA at the time of the first vaccination.
5. Healthy subjects as established by medical history and clinical examination before entering into the study.
6. Female subjects of non-childbearing potential may be enrolled in the study.

   * Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
7. Female subjects of childbearing potential may be enrolled in the study, if the subject:

   * has practiced adequate contraception for 30 days prior to vaccination, and
   * has a negative pregnancy test on the day of vaccination, and
   * has agreed to continue adequate contraception during the entire treatment period. (approximately 1 month after vaccination).

Exclusion Criteria:

1. Anaphylaxis following the administration of vaccine
2. Any (clinical) condition that in the judgment of the investigator would make intramuscular injection unsafe and/or represents a contraindication to intramuscular vaccination and blood draws.
3. Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection.
4. Progressive, unstable or uncontrolled clinical conditions.
5. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
6. Hypersensitivity to the active substances or to any of the excipients of the vaccine, including diphtheria toxoid (CRM197), or a life-threatening reaction after previous administration of a vaccine containing similar components.
7. Abnormal function of the immune system resulting from:

   * Clinical conditions.
   * Systemic administration of corticosteroids (Per os [PO]/ Intravenous [IV]/ Intramuscular [IM]) for more than 14 consecutive days within 90 days prior to informed consent, and until the Day 29 blood draw.
   * Administration of antineoplastic and immuno-modulating agents or radiotherapy within 90 days prior to informed consent, and until the Day 29 blood draw.
8. Received immunoglobulins or any blood products within 180 days prior to informed consent.
9. Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
10. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
11. History of any meningococcal vaccination.
12. Individuals who received any other vaccines within 7 days (for inactivated vaccines) or 14 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccines*.

    * In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its Summary of Product Characteristics (SmPC) or Prescribing Information and according to the local governmental recommendations and provided a written approval of the Sponsor is obtained.
13. Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
14. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product. (pharmaceutical product or device).
15. Current or previous, confirmed or suspected disease caused by N. meningitidis.
16. Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days prior to study vaccination.
17. Acute disease and/or fever within 3 days prior to study vaccination. Note: enrolment may be postponed/delayed until such transient circumstances have ended.

    * Fever is defined as body temperature ≥ 38.0°C / 100.4°F. The preferred location for measuring temperature in this study will be the oral cavity.
    * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
18. Received systemic antibiotic treatment within 3 days prior to study vaccination or blood draw.
19. Study personnel as an immediate family or household member.
20. Pregnant or lactating women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 996 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- Australia (8):
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Kanwal, New South Wales
  - GSK Investigational Site, Gold Coast, Queensland
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
  - GSK Investigational Site, Melbourne
- Belgium (2):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Canada (10):
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Germany (6):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (4):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Conegliano - Treviso
  - GSK Investigational Site, Massafra (TA)

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Vir Singh P, Tiberi P, Di Domenico GF, Romolini V, Mzolo T, Costantini M, Akhund T, Basile V, Lattanzi M, Pellegrini M. Fully Liquid MenACWY-CRM Vaccine: Results from an Integrated Safety Analysis. Drug Saf. 2023 Jan;46(1):99-108. doi: 10.1007/s40264-022-01242-8. Epub 2022 Nov 11. PMID 36369456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 8 centers in Australia, 2 in Belgium, 10 in Canada, 6 in Germany and 4 in Italy.Planned age range in this study was 18-40 years.But 1 subject aged 44 years not meeting inclusion criteria was enrolled & vaccinated in GSK3536820A ACWY_Liq Group & therefore was considered for all analyses except per protocol set for immunogenicity analyses
Pre-assignment Details: Among 996 enrolled subjects, 16 subjects didn't receive any treatment and ICF documentation was not retrievable for 1 subject.
Groups:
- GSK3536820A ACWY_Liq Group: Healthy adults, 18 to 44 years of age, receiving at Day 1 a single dose of investigational MenACWY liquid vaccine (GSK3536820A) formulation with approximately 30% Men A FS.
- ACWY Group: Healthy adults, 18 to 40 years of age, receiving at Day 1 a single dose of licensed GSK's MenACWY vaccine formulation (Menveo).
Period: Overall Study
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Started | 490 | 489
Completed | 486 | 484
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group | Total
Number analyzed (Participants) | 490 | 489 | 979
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (5.8) | 31.9 (5.8) | 31.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 309 | 305 | 614
  Male | 181 | 184 | 365
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 4 | 0 | 4
  Asian | 40 | 27 | 67
  Black Or African American | 4 | 8 | 12
  Native Hawaiian Or Other Pacific Islander | 2 | 2 | 4
  Other | 13 | 13 | 26
  White | 427 | 439 | 866

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Human Serum Bactericidal Activity (hSBA) Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroup A for Each Vaccine Group, and Between-group Ratios
Description: hSBA titers against N.meningitidis serogroup A were calculated in terms of GMTs adjusted for pre-vaccination titer.
Time Frame: At Day 29
Population: Analysis was performed on the per protocol set for immunogenicity that includes subjects who received the vaccine, did not have any protocol deviation leading to exclusion, who were not excluded due to other reasons defined prior to unblinding or analysis and had available immuno data for any serogroup and time point considered.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 386 | 404
Titers | 185.16 [147.90 to 231.81] | 211.33 [169.61 to 263.32]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; To demonstrate non-inferiority of the investigational MenACWY liquid vaccine with approximately 30% Men A FS (GSK3536820A ACWY_Liq Group) to that of currently licensed MenACWY vaccine (ACWY Group), as measured by the adjusted human serum bactericidal assay (hSBA) Geometric Mean Titers (GMTs) directed against N. meningitidis serogroup A at Day 29 after a single dose vaccination; Test type: Non-Inferiority — Non-inferiority is concluded if the lower limit of the two sided 95% CI for the hSBA GMT ratio for serogroup A is > 0.5; ANCOVA; Analysis of Covariance (ANCOVA) including pre-vaccination titer (Day 1) as a covariate and with vaccine group and country as factors; GMT ratio = 0.88, 95% CI 2-sided [0.64 to 1.20]

2. Secondary Outcome: hSBA GMTs Against Each of the N.Meningitidis Serogroups A, C, W and Y for Each Vaccine Group, and Between-group Ratios
Description: hSBA titers were calculated in terms of GMTs, at Day 1 and Day 29, against each of the N. meningitidis serogroups A, C, W and Y.
Time Frame: At Day 1 and Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 459 | 467
Titers
  Meningitis A, Day 1: number analyzed (Participants) | 446 | 446
  Meningitis A, Day 1 | 2.79 [2.52 to 3.10] | 2.97 [2.68 to 3.29]
  Meningitis A, Day 29: number analyzed (Participants) | 386 | 404
  Meningitis A, Day 29 | 182.96 [145.11 to 230.68] | 213.42 [170.11 to 267.77]
  Meningitis C, Day 1 | 11.41 [9.81 to 13.27] | 12.05 [10.38 to 14.00]
  Meningitis C, Day 29: number analyzed (Participants) | 437 | 441
  Meningitis C, Day 29 | 153.95 [115.03 to 206.04] | 139.63 [104.56 to 186.47]
  Meningitis W, Day 1: number analyzed (Participants) | 455 | 457
  Meningitis W, Day 1 | 9.6 [8.05 to 11.45] | 10.92 [9.16 to 13.02]
  Meningitis W, Day 29: number analyzed (Participants) | 445 | 443
  Meningitis W, Day 29 | 59.74 [47.67 to 74.86] | 54.12 [43.17 to 67.86]
  Meningitis Y, Day 1: number analyzed (Participants) | 458 | 463
  Meningitis Y, Day 1 | 4.14 [3.63 to 4.71] | 4.75 [4.17 to 5.40]
  Meningitis Y, Day 29: number analyzed (Participants) | 452 | 455
  Meningitis Y, Day 29 | 60.29 [48.67 to 74.68] | 54.99 [44.44 to 68.06]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; To compare the immunogenicity of the investigational MenACWY liquid vaccine with approximately 30% Men A FS (GSK3536820A ACWY_Liq Group) and the currently licensed MenACWY vaccine (ACWY Group), as measured by the adjusted hSBA GMTs directed against N. meningitidis serogroup C at Day 29; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.19, 95% CI 2-sided [0.84 to 1.68]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; To compare the immunogenicity of the investigational MenACWY liquid vaccine with approximately 30% Men A FS (GSK3536820A ACWY_Liq Group) and the currently licensed MenACWY vaccine (ACWY Group), as measured by the adjusted hSBA GMTs directed against N. meningitidis serogroup W at Day 29; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.23, 95% CI 2-sided [0.96 to 1.58]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; To compare the immunogenicity of the investigational MenACWY liquid vaccine with approximately 30% Men A FS (GSK3536820A ACWY_Liq Group) and the currently licensed MenACWY vaccine (ACWY Group), as measured by the adjusted hSBA GMTs directed against N. meningitidis serogroup Y at Day 29; Test type: Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; GMT ratio = 1.19, 95% CI 2-sided [0.90 to 1.58]

3. Secondary Outcome: Within-group Geometric Mean Ratios (GMRs) Against Each of the N.Meningitidis Serogroups A, C, W and Y
Description: Within-group ratios of hSBA GMTs against each of the N.meningitidis serogroups A, C, W and Y at Day 29 compared to Day 1.
Time Frame: At Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 452 | 455
Ratio
  Meningitis A: number analyzed (Participants) | 386 | 404
  Meningitis A | 65.24 [51.81 to 82.16] | 73.01 [58.26 to 91.49]
  Meningitis C: number analyzed (Participants) | 437 | 441
  Meningitis C | 13.17 [10.30 to 16.84] | 11.07 [8.68 to 14.13]
  Meningitis W: number analyzed (Participants) | 445 | 443
  Meningitis W | 6.1 [5.07 to 7.33] | 4.8 [3.99 to 5.77]
  Meningitis Y | 14.64 [11.88 to 18.04] | 11.48 [9.33 to 14.13]

4. Secondary Outcome: Percentages of Subjects With a ≥4 Fold Rise in hSBA Antibody Titers for Each of the N.Meningitidis Serogroups A, C,W and Y for Each Vaccine Group, and Between-group Differences
Description: The percentages of subjects with a ≥ 4-fold rise in post-vaccination hSBA (at Day 29 compared to Day 1) and associated 2-sided 95% Clopper-Pearson CIs were computed by group and for each N. meningitidis serogroups A, C, W and Y. A 4-fold rise in the hSBA titers is defined as: for individuals, whose pre-vaccination titers are < the LOD (limit of detection), the post-vaccination titers must be ≥ 4-fold the LOD or ≥ the LLOQ (lower of limit of quantitation) whichever is greater; for individuals, whose pre-vaccination titers are ≥ the LOD and ≤ the LLOQ, the post-vaccination titers must be at least four times the LLOQ; for individuals whose pre-vaccination titers are > the LLOQ, the post-vaccination titers must be at least four times the pre-vaccination
Time Frame: At Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 452 | 455
Percentages of subjects
  Meningitis A: number analyzed (Participants) | 386 | 404
  Meningitis A | 79.8 [75.4 to 83.7] | 83.7 [79.7 to 87.1]
  Meningitis C: number analyzed (Participants) | 437 | 441
  Meningitis C | 56.3 [51.5 to 61.0] | 54.4 [49.6 to 59.1]
  Meningitis W: number analyzed (Participants) | 445 | 443
  Meningitis W | 44.7 [40.0 to 49.5] | 40.2 [35.6 to 44.9]
  Meningitis Y | 63.3 [58.6 to 67.7] | 58 [53.3 to 62.6]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup A at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -3.87, 95% CI 2-sided [-9.30 to 1.52]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup C at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.87, 95% CI 2-sided [-4.70 to 8.43]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup W at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 4.54, 95% CI 2-sided [-1.97 to 11.01]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentage of subjects with a ≥ 4-fold rise in post-vaccination hSBA for N. meningitidis serogroup Y at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 5.25, 95% CI 2-sided [-1.11 to 11.57]

5. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥8 Against Each of the N. Meningitidis Serogroups A, C, W and Y for Each Vaccine Group, and Between-group Differences
Description: For each vaccine group the percentage of subjects with hSBA titer ≥8, and its associated two-sided 95% Clopper-Pearson CIs were computed for each of the N. meningitidis serogroups A, C, W and Y.
Time Frame: At Day 1 and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 460 | 467
Percentages of subjects
  Meningitis A, Day 1: number analyzed (Participants) | 446 | 446
  Meningitis A, Day 1 | 8.7 [6.3 to 11.8] | 11.2 [8.4 to 14.5]
  Meningitis A, Day 29: number analyzed (Participants) | 406 | 428
  Meningitis A, Day 29 | 82.8 [78.7 to 86.3] | 86.4 [82.8 to 89.5]
  Meningitis C, Day 1: number analyzed (Participants) | 459 | 467
  Meningitis C, Day 1 | 53.8 [49.1 to 58.4] | 54.4 [49.7 to 59.0]
  Meningitis C, Day 29: number analyzed (Participants) | 443 | 446
  Meningitis C, Day 29 | 74.5 [70.2 to 78.5] | 74.9 [70.6 to 78.8]
  Meningitis W, Day 1: number analyzed (Participants) | 455 | 457
  Meningitis W, Day 1 | 39.8 [35.3 to 44.4] | 45.7 [41.1 to 50.4]
  Meningitis W, Day 29: number analyzed (Participants) | 454 | 457
  Meningitis W, Day 29 | 73.3 [69.0 to 77.4] | 73.1 [68.8 to 77.1]
  Meningitis Y, Day 1: number analyzed (Participants) | 458 | 463
  Meningitis Y, Day 1 | 22.7 [18.9 to 26.8] | 25.5 [21.6 to 29.7]
  Meningitis Y, Day 29: number analyzed (Participants) | 460 | 463
  Meningitis Y, Day 29 | 77.2 [73.1 to 80.9] | 76 [71.9 to 79.8]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup A at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -2.47, 95% CI 2-sided [-6.47 to 1.49]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup C at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.58, 95% CI 2-sided [-6.99 to 5.83]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup W at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -5.95, 95% CI 2-sided [-12.33 to 0.47]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup Y at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -2.78, 95% CI 2-sided [-8.30 to 2.76]
Statistical Analysis 5: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup A at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -3.69, 95% CI 2-sided [-8.65 to 1.21]
Statistical Analysis 6: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup C at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.40, 95% CI 2-sided [-6.12 to 5.33]
Statistical Analysis 7: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup W at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.26, 95% CI 2-sided [-5.49 to 6.02]
Statistical Analysis 8: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥8 for the N. meningitidis serogroup Y at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 1.15, 95% CI 2-sided [-4.33 to 6.62]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLOQ Against Each of the N. Meningitidis Serogroups A, C, W and Y for Each Vaccine Group, and Between-group Differences
Description: For each vaccine group the percentage of subjects with hSBA titer ≥LLOQ, and its associated two-sided 95% Clopper-Pearson CIs were computed for each of the N. meningitidis serogroups A, C, W and Y.
Time Frame: At Day 1 and Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 460 | 467
Percentages of subjects
  Meningitis A, Day 1: number analyzed (Participants) | 446 | 446
  Meningitis A, Day 1 | 10.5 [7.8 to 13.8] | 13.5 [10.4 to 17.0]
  Meningitis A, Day 29: number analyzed (Participants) | 406 | 428
  Meningitis A, Day 29 | 82.8 [78.7 to 86.3] | 86.7 [83.1 to 89.8]
  Meningitis C, Day 1: number analyzed (Participants) | 459 | 467
  Meningitis C, Day 1 | 61.2 [56.6 to 65.7] | 62.3 [57.7 to 66.7]
  Meningitis C, Day 29: number analyzed (Participants) | 443 | 446
  Meningitis C, Day 29 | 76.5 [72.3 to 80.4] | 76.5 [72.2 to 80.3]
  Meningitis W, Day 1: number analyzed (Participants) | 455 | 457
  Meningitis W, Day 1 | 41.3 [36.8 to 46.0] | 47.3 [42.6 to 52.0]
  Meningitis W, Day 29: number analyzed (Participants) | 454 | 457
  Meningitis W, Day 29 | 73.3 [69.0 to 77.4] | 73.5 [69.2 to 77.5]
  Meningitis Y, Day 1: number analyzed (Participants) | 458 | 463
  Meningitis Y, Day 1 | 23.8 [20.0 to 28.0] | 26.3 [22.4 to 30.6]
  Meningitis Y, Day 29: number analyzed (Participants) | 460 | 463
  Meningitis Y, Day 29 | 77.8 [73.7 to 81.5] | 77.3 [73.2 to 81.1]
Statistical Analysis 1: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup A at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -2.91, 95% CI 2-sided [-7.24 to 1.37]
Statistical Analysis 2: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup C at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -1.09, 95% CI 2-sided [-7.34 to 5.16]
Statistical Analysis 3: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup W at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -5.95, 95% CI 2-sided [-12.35 to 0.50]
Statistical Analysis 4: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup Y at Day 1; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -2.55, 95% CI 2-sided [-8.15 to 3.06]
Statistical Analysis 5: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup A at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -3.92, 95% CI 2-sided [-8.87 to 0.96]
Statistical Analysis 6: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup C at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.07, 95% CI 2-sided [-5.52 to 5.65]
Statistical Analysis 7: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup W at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = -0.17, 95% CI 2-sided [-5.92 to 5.57]
Statistical Analysis 8: Comparison: GSK3536820A ACWY_Liq Group vs ACWY Group; Between-group difference in percentages of subjects with hSBA titer ≥LLOQ for the N. meningitidis serogroup Y at Day 29; Test type: Other; Miettinen and Nurminen score method; Difference in percentage of subjects = 0.50, 95% CI 2-sided [-4.89 to 5.90]

7. Secondary Outcome: Number of Subjects Reported With Solicited Local and Systemic AEs
Description: Number of subjects with solicited local and systemic AEs during the 7-days period (including the day of vaccination) after the vaccination.
Time Frame: From Day 1 (6 hours) to Day 7 after vaccination
Population: Analysis was performed on the solicited safety set that includes all enrolled subjects who received a study vaccination and reported any solicited adverse events data for the defined period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 489 | 487
Participants
  Erythema | 28 | 28
  Induration | 25 | 24
  Pain | 200 | 182
  Arthralgia | 43 | 46
  Chills | 42 | 40
  Fatigue | 159 | 159
  Fever (Temperature >= 38 C) | 7 | 10
  Headache | 158 | 165
  Loss of Appetite | 31 | 40
  Myalgia | 58 | 58
  Nausea | 49 | 50

8. Secondary Outcome: Number of Subjects Reported With Other Indicators of Reactogenicity
Description: Number of subjects reporting other indicators of reactogenicity such as use of analgesics/antipyretics within 7 days after vaccination
Time Frame: From Day 1 to Day 7 after vaccination
Population: Analysis was performed on the solicited safety set that includes all enrolled subjects who received a study vaccination and reported any indicators of reactogenicity data for the defined period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 489 | 487
Participants
  Analgesic/Antipyretic Prevention, Yes | 36 | 40
  Analgesic/Antipyretic Prevention, No | 453 | 447
  Analgesic/Antipyretic Treatment, Yes | 80 | 79
  Analgesic/Antipyretic Treatment, No | 409 | 408

9. Secondary Outcome: Number of Subjects Reported With Any Unsolicited AEs Within 29 Days After Vaccination
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered with a pharmaceutical product at any dose that does not necessarily have to have a causal relationship with this treatment.
Time Frame: From Day 1 to Day 29 after vaccination
Population: Analysis was performed on the unsolicited safety set that includes all enrolled subjects who received a study vaccination and reported unsolicited adverse events data for the defined period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 489 | 489
Participants | 117 | 111

10. Secondary Outcome: Number of Subjects Reported With AEs Leading to Withdrawal, Medically Attended AEs and Serious Adverse Events (SAEs)
Description: Medically attended AEs are defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any medically attended AE(s) is occurrence of any medically attended AE(s) regardless of intensity grade or relation to vaccination. Serious adverse event is any congenital anomaly/birth defect in the offspring of a study subject or any untoward medical occurrence that results in death or life threatening or requires hospitalization or results in disability or incapacity
Time Frame: From Day 1 to Day 181 (during the entire study period)
Population: Analysis was performed on the unsolicited safety set that includes all enrolled subjects who received a study vaccination and reported any adverse events data in the defined period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 489 | 489
Participants
  Aes leading to withdrawal | 0 | 0
  MAEs | 79 | 84
  SAEs | 6 | 9

11. Secondary Outcome: Number of Subjects Reported With Any Unsolicited Adverse Events (AEs) Within 30 Minutes After Vaccination
Description: as for outcome 9
Time Frame: Within 30 minutes after vaccination at Day 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
Number analyzed (Participants) | 489 | 489
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7 after vaccination and Unsolicited AEs from Day 1 to Day 29 after vaccination. SAEs were collected from Day 1 to Day 181 (during the entire study period)
Arm/Group | GSK3536820A ACWY_Liq Group | ACWY Group
All-Cause Mortality (participants affected / at risk) | 0/490 | 0/489
Serious Adverse Events (participants affected / at risk) | 6/490 | 9/489
Other Adverse Events (participants affected / at risk) | 336/490 | 335/489
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3536820A ACWY_Liq Group (N=490) | ACWY Group (N=489)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3536820A ACWY_Liq Group (N=490) | ACWY Group (N=489)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 51 (52) | 51 (52)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Administration site joint pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 43 (44) | 40 (40)
Fatigue (General disorders) | 160 (163) | 162 (163)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 5 (5) | 2 (2)
Injection site bruising (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 30 (31) | 31 (32)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 26 (27) | 25 (25)
Injection site joint pain (General disorders) | 1 (2) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 200 (204) | 184 (184)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 1 (1)
Injection site warmth (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 10 (11) | 10 (10)
Vaccination site induration (General disorders) | 1 (1) | 0 (0)
Vaccination site paraesthesia (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Candida infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 11 (11) | 10 (10)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 6 (6)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Streptococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 31 (31) | 41 (42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 (44) | 49 (49)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 59 (59) | 58 (58)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 162 (167) | 171 (183)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT03652610/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03652610/SAP_001.pdf